CLINICAL TRIAL: NCT01548794
Title: A Comparison of the Recovery Profiles of Bupivacaine or Bupivacaine Mixed With Lidocaine Spinal Anesthesia and Local Infiltration Anesthesia for Outpatient Herniorrhaphy
Brief Title: Recovery of Bupivacaine or Bupivacaine-Lidocaine Spinal Anesthesia and Infiltration Anesthesia in Herniorrhaphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Doctor Specialist in Anesthesiology Principal investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DiskapiTRHDYAZICIOGLU
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2012-12

CONDITIONS: Anesthesia; Inguinal Hernia
Keywords: spinal anesthesia; bupivacaine; lidocaine; local infiltration anesthesia; recovery; duration of anesthesia; outpatient herniorrhaphy
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Spinal; Lidocaine; Anesthesia, Local; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bupivacaine(Group B) (Active Comparator): spinal anesthesia
  Interventions: Procedure: spinal anesthesia
- Bupivacaine+Lidocaine (Group BL) (Experimental): spinal anesthesia
  Interventions: Procedure: spinal anesthesia
- Local Infitration Anesthesia(Group LI) (Active Comparator): local infiltration anesthesia
  Interventions: Procedure: infiltration anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — To receive 2 ml heavy bupivacaine + 0,6 ml saline
  Other Names: marcaine heavy
  Arms: Bupivacaine(Group B)
Procedure: spinal anesthesia — To receive 2ml bupivacaine +0,6 ml 1% lidocaine for spinal anesthesia.
  Other Names: marcaine heavy; lidocaine
  Arms: Bupivacaine+Lidocaine (Group BL)
Procedure: infiltration anesthesia — To receive step by step local infiltration anesthesia as described by the Lichtenstein Institute.
  Other Names: marcaine; lidocaine
  Arms: Local Infitration Anesthesia(Group LI)

SUMMARY:
The purpose of this study is the investigation of whether adding lidocaine to hyperbaric bupivacaine could decrease the duration of bupivacaine spinal block and provide shorter recovery and discharge times than local infiltration anesthesia in outpatient herniorrhaphy procedures.

DETAILED DESCRIPTION:
Consecutive 93 patients undergoing inguinal herniorrhaphy will be recruited with a prospective protocol.Spinal anesthesia will be commenced in Group BLS with 2 ml hyperbaric bupivacaine (10 mg) + 0.6 ml 1 % lidocaine (6 mg), in Group BS, hyperbaric bupivacaine (10 mg) + saline in the same volume and Group LIA will have anesthesia with bupivacaine and lidocaine for step by step local anesthetic infiltration. Sensorial block will be measured with pinprick test, motor block will be tested with Bromage scale. Heart rate, blood pressure and peripheral oxygen saturation will be measured every 5 minutes. Time of subarachnoid injection, onset of sensorial block (block at L1 dermatome), time to block T10 dermatome, maximum block level, time to maximum block and time to two segment regression, T10 regression , LI regression and S1 regression of the block will be recorded in group BLS and BS.The onset and resolution of the sensorial and motor block will be assessed by anesthetists blinded to group allocation. PACU stay and discharge times and VAS pain scores will be recorded in all patients. Patients also will be investigated for adverse events (hypotension, bradycardia, nausea,PDPH, TNS, urinary retention)and satisfaction regarding the anesthetic method.

ELIGIBILITY:
Inclusion Criteria:

* Patients having inguinal hernia
* Not hypersensitive to study drugs
* ASA classification I-III

Exclusion Criteria:

* ASA classification IV-V
* Contraindications for spinal anesthesia

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Duration of spinal block | day of surgery
  Time between the onset of the sensorial block at L1 dermatome and the resolution of the sensorial block at S3 dermatome.

SECONDARY OUTCOMES:
Discharge time | Day of surgery
  The time between the end of surgery and home discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yazicioglu, Principal Investigator
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Lee SJ, Bai SJ, Lee JS, Kim WO, Shin YS, Lee KY. The duration of intrathecal bupivacaine mixed with lidocaine. Anesth Analg. 2008 Sep;107(3):824-7. doi: 10.1213/ane.0b013e3181806149. PMID 18713891